CLINICAL TRIAL: NCT00325065
Title: Identifying the Role of Oxytocin and Vasopressin in the Functioning of Neurocognitive Systems Involved in Mood Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060155; 06-M-0155
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-04-16

CONDITIONS: Mood Disorders
Keywords: Amygdala; Emotion; Memory; Threat; Peptides; Neuropeptides; Oxytocin; Vasopressin; Mood Disorder
MeSH Terms: conditions — Mood Disorders; Diabetes Insipidus

SUMMARY:
The goal of this protocol, broadly stated, is to use targeted manipulations with intranasally administered oxytocin (OT) and arginine vasopressin (AVP) in conjunction with neurocognitive and neuroimaging paradigms to evaluate claims that OT and AVP inhibit and facilitate, respectively, the effective processing of aversive signals. Moreover, we wish to examine whether increased vasopressin levels will increase, and increased oxytocin levels decrease, the neural response in the amygdala and other limbic structures to aversive stimuli. In addition, we wish to assess whether OT and AVP administration will lead to the facilitation of conspecific recognition as appears to be the case for other mammalian species....

DETAILED DESCRIPTION:
Objective:

The goal of this protocol, broadly stated, is to use targeted manipulations with intranasally administered oxytocin (OT) and arginine vasopressin (AVP) in conjunction with neurocognitive and neuroimaging paradigms to evaluate claims that OT and AVP inhibit and facilitate, respectively, the effective processing of aversive signals.

Study Population:

A total of 216 healthy male and female adults between 20-40 years of age.

Design:

This protocol will involve a series of independent studies. Each study will require one visit in addition to a screening visit, involves a physical and psychiatric assessment. The study visit itself will involve pharmacological challenge followed by neurocognitive or neuroimaging testing.

Outcome Measures:

Moreover, we wish to examine whether increased vasopressin levels will increase, and increased oxytocin levels decrease, the neural response in the amygdala and other limbic structures to aversive stimuli. In addition, we wish to assess whether OT and AVP administration will lead to the facilitation of conspecific recognition as appears to be the case for other mammalian species.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age: Participants will be healthy males and females, 20-40 years of age. Approximately equal numbers of males and females will be included in each study.
  2. IQ: IQ, as measured by 4 subscales from the Wechsler Adult Intelligence Scale-Revised (WAIS-R), must be greater than 80. Prior testing in our laboratory has indicated that this cutoff allows for maximally generalizeable results while ensuring that all participants will understand and be able to complete the testing procedures.
  3. Menstrual phase: Female participants will be tested only during the follicular phase of their menstrual cycle (defined as days 6-12 after the first day of the last menstrual period and confirmed using ovulation testing kits).

EXCLUSION CRITERIA:

Because factors such as psychiatric disease or CNS disease can influence functional brain activity, these factors are exclusionary.

1. Psychiatric history: Participants will be assessed using DSM-IV criteria via standardized psychiatric interviews conducted by trained examiners (SCID). All participants will be free of any current or past major affective disorder, psychotic disorder, substance dependence, anorexia, somatoform disorder, or anxiety disorders including specific phobias.
2. Medical Illnesses: Moderate or severe acute or chronic medical illnesses (e.g. cardiac disease, diabetes, epilepsy, influenza).
3. Cardiovascular risk factors: History of hypertension with baseline blood pressure above 140 mm Hg (systolic) over 85 mm Hg (diastolic). Also any history of syncope and/or baseline blood pressure below 100 mm Hg (systolic).
4. CNS disease: Known history of brain abnormalities (e.g., neoplasms, subarachnoid cysts), cerebrovascular disease, infectious disease (e.g., abscess), other central nervous system disease, or history of head trauma which resulted in a persistent neurologic deficit or loss of consciousness greater than 3 minutes.
5. Medication status: Currently on regular medication that would interfere with study results. This includes contraceptive hormones, psychotropic medications or benzodiazepines, alpha and beta adrenergic medications, other anti-hypertensive medications, glucocorticoid and mineralocorticoid medications, and medications causing sedation or stimulation. For example, current use of acetaminophen or ibuprofen is permitted, while current use of benadryl or methylphenidate is not.
6. Pregnancy or Nursing Status: Currently breast feeding or pregnant (as documented by pregnancy testing which will be performed at screening and on the day of the challenge study).

ADDITIONAL EXCLUSION CRITERIA FOR FMRI STUDIES:

1. Metal or electronic objects: Metal plates, certain types of dental braces, cardiac pacemakers, etc., that are sensitive to electromagnetic fields contraindicate MRI scans.
2. Claustrophobia: Participants will be questioned about potential discomfort in being in an enclosed space, such as an MRI scanner.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2006-05-05; Study Completion 2010-04-16

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bohus B, Kovacs GL, de Wied D. Oxytocin, vasopressin and memory: opposite effects on consolidation and retrieval processes. Brain Res. 1978 Nov 24;157(2):414-7. doi: 10.1016/0006-8993(78)90052-5. No abstract available. PMID 719533
- [Background] DeVries AC, Glasper ER, Detillion CE. Social modulation of stress responses. Physiol Behav. 2003 Aug;79(3):399-407. doi: 10.1016/s0031-9384(03)00152-5. PMID 12954434
- [Background] Dyball RE, Paterson AT. Neurohypophysial hormones and brain function: the neurophysiological effects of oxytocin and vasopressin. Pharmacol Ther. 1983;20(3):419-36. doi: 10.1016/0163-7258(83)90035-9. PMID 6136996